CLINICAL TRIAL: NCT00018486
Title: Epidemiology of Hearing Loss in Diabetic and Non-Diabetic Veterans
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: EPID-018-98F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Diabetes; Tinnitus; Hearing Loss
MeSH Terms: conditions — Diabetes Mellitus; Tinnitus; Hearing Loss

SUMMARY:
The purpose of this study is to determine if individuals with diabetes are at increased risk of hearing impairment or tinnitus (the perception of ringing or noises in the ears or head). An important goal of this research is also to obtain a better understanding of possible interactions between hearing disorders and other chronic conditions, such as diabetes. Participation in this research will be for a few hours only, to be scheduled at the participant's convenience and according to the testing schedules of the different clinics involved.

ELIGIBILITY:
Any participants over 21 years of age and under 80 who do not have an end-stage disease

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1999-04; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (1):
- Portland VA Medical Center, Portland, Oregon, United States